CLINICAL TRIAL: NCT00966927
Title: Assessment of Functional Independence and Quality of Life in Italian Population of Adolescents With Spina Bifid
Brief Title: Assessment of Functional Independence and Quality of Life in Adolescents With Spina Bifid
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: UDGEE-SPINA BIFIDA
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Spinal Dysraphism
Keywords: quality of life; functional independence; spina bifid
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subjects with spina bifid: subjects with spina bifid between 14 and 21 years old referred to Unit for Care of Spina Bifid Hospital of Parma

SUMMARY:
The purpose of this study is to investigate the level of functional independence and the quality of life of adolescents and young adults with spina bifid in an Italian population.

DETAILED DESCRIPTION:
We submitted the Quality of Life in spina bifid Questionnaire to subjects who participated in the study and the Spinal Cord Independence Measure to the parents of subjects.

ELIGIBILITY:
Inclusion Criteria:

* recurrence of clinic control in Unit for Spina Bifid in Parma
* 14-21 years old

Exclusion Criteria:

* subjects unable to understand the items of the questionnaire (mental retardation and need for help at school )
* subjects without any caregiver

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: subjects with spina bifid referred to primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
correlation between the quality of life in adolescents and young adults with Spina Bifid and their level of functional independence | 5 months

SECONDARY OUTCOMES:
correlation between functional level of independence and motor level of neurological lesion | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Care of Spina Bifida, Parma, Parma, Italy

REFERENCES:
- [Background] Buran CF, Sawin KJ, Brei TJ, Fastenau PS. Adolescents with myelomeningocele: activities, beliefs, expectations, and perceptions. Dev Med Child Neurol. 2004 Apr;46(4):244-52. doi: 10.1017/s0012162204000404. PMID 15077702